CLINICAL TRIAL: NCT07389278
Title: A Phase 1/2 Study of Pegylated Arginine Deiminase (ADI-PEG 20) Plus Radiotherapy (RT) and Temozolomide (TMZ) in Children, Adolescents, and Young Adults With Newly Diagnosed High-grade Glioma (HGG)
Brief Title: Combination ADI-PEG 20, TMZ, and RT for Treatment of Newly Diagnosed High-grade Glioma (HGG)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 250814; NCI-2026-00045 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; High-Grade Glioma (WHO III-IV); High-grade Glioma; Diffuse Midline Glioma, H3 K27M-Mutant; Diffuse Hemispheric Glioma, H3G34 Mutant
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — ADI PEG20; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 (Starting Dose: ADI-PEG 20 36mg/m^2) (Experimental): Participants will receive injection of 36 mg/m^2 of ADI-PEG 20 once weekly in the concomitant phase and maintenance phases given prior to the start of RT. Participants will also receive daily oral (PO) temozolomide (TMZ) with dosage based on age and dosing phase (concomitant, then maintenance) starting on the same day as Radiotherapy (RT). RT will be given in standard fractions (total dose 59.4 Gy) over 6 weeks. The boost volume, when present, will receive an additional 5.4 Gy for a total of 59.4 Gy. Post-RT, Participants will continue to receive weekly ADI-PEG 20 as monotherapy and then proceed to first cycle of maintenance therapy 28 days (+7 days) after completion of RT, in the absence of dose-limiting toxicities (DLT) or progressive disease. The maintenance phase consists of ten cycles (28 days long) of combination chemotherapy with ADI-PEG 20 and TMZ. Participants will receive no more than 104 weeks of ADI-PEG 20 therapy
  Interventions: Drug: Temozolomide (TMZ); Radiation: Standard of Care Radiation Therapy (RT)
- Phase 2 (Cohort 1) - Histone Wild Type (WT) HGG (Experimental): Participants with WT HGG will be treated at the recommended phase 2 dose (RP2D) of ADI-PEG 20 determined in Phase 1 in combination with TMZ. Participants who complete the combined treatment and maintenance phase may continue receiving monotherapy treatment as extended maintenance for up to 10 additional cycles, provided there is no unacceptable toxicity, disease progression, or withdrawal of consent. ADI-PEG 20 treatment may continue for up to 104 weeks.
  Interventions: Drug: ADI-PEG 20 (Arginine deiminase pegylated); Drug: Temozolomide (TMZ); Radiation: Standard of Care Radiation Therapy (RT)
- Phase 2 (Cohort 2) - H3K27 Altered Diffuse Midline Gliomas (DMG) (Experimental): Participants will be treated at the recommended phase 2 dose (RP2D) of ADI-PEG 20 determined in Phase 1. Participants who complete the combined treatment and maintenance phase may continue receiving monotherapy treatment as extended maintenance for up to 10 additional cycles, provided there is no unacceptable toxicity, disease progression, or withdrawal of consent. ADI-PEG 20 treatment may continue for up to 104 weeks. After completing the 30-day toxicity evaluation period, participants will enter follow-up. Follow-up procedures will be documented under the PNOC COMP protocol, except for protocol-defined follow-up procedures. Participants will be followed under the PNOC COMP protocol until death or withdrawal from the study.
  Interventions: Drug: ADI-PEG 20 (Arginine deiminase pegylated); Drug: Temozolomide (TMZ); Radiation: Standard of Care Radiation Therapy (RT)
- Phase 2 (Cohort 3) - H3G34 Mutant Diffuse Hemispheric Gliomas (DHG) (Experimental): Participants will be treated at the recommended phase 2 dose (RP2D) of ADI-PEG 20 determined in Phase 1. Participants who complete the combined treatment and maintenance phase may continue receiving monotherapy treatment as extended maintenance for up to 10 additional cycles, provided there is no unacceptable toxicity, disease progression, or withdrawal of consent. ADI-PEG 20 treatment may continue for up to 104 weeks. After completing the 30-day toxicity evaluation period, participants will enter follow-up. Follow-up procedures will be documented under the PNOC COMP protocol, except for protocol-defined follow-up procedures. Participants will be followed under the PNOC COMP protocol until death or withdrawal from the study.
  Interventions: Drug: ADI-PEG 20 (Arginine deiminase pegylated); Drug: Temozolomide (TMZ); Radiation: Standard of Care Radiation Therapy (RT)

INTERVENTIONS:
Drug: ADI-PEG 20 (Arginine deiminase pegylated) — Given intramuscularly (IM)
  Other Names: ADI-PEG 20
  Arms: Phase 2 (Cohort 1) - Histone Wild Type (WT) HGG; Phase 2 (Cohort 2) - H3K27 Altered Diffuse Midline Gliomas (DMG); Phase 2 (Cohort 3) - H3G34 Mutant Diffuse Hemispheric Gliomas (DHG)
Drug: Temozolomide (TMZ) — Given orally (PO)
  Other Names: TMZ
Radiation: Standard of Care Radiation Therapy (RT) — Undergo RT
  Other Names: RT

SUMMARY:
This is an open label, intra-patient dose escalation, to evaluate ADI-PEG 20, in combination with Temozolomide (TMZ) and radiation therapy (RT) in children, adolescents and young adult patients with newly diagnosed high grade glioma (HGG).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and estimate the RP2D of ADI-PEG 20 in combination with RT and TMZ in with children, adolescents, and young adults with newly diagnosed high-grade glioma, and the RP2D of ADI-PEG 20 during maintenance therapy with TMZ (Phase 1)

II. To assess the anti-tumor activity of the combination of ADI-PEG 20 with RT and TMZ based on progression-free survival (PFS) at 12 months for HGG histone-WT participants, 12 months for H3K27 altered DMG, and 10 months for H3G34 mutant DHG in children, adolescents, and young adult participants (Phase 2)

EXPLORATORY OBJECTIVES:

I. To assess the anti-tumor activity of the combination of ADI-PEG 20 with RT and TMZ based on overall survival at 12 months for HGG histone-WT, Histone 3 lysine 27 (H3K27) altered DMG, and Histone 3 G34-mutant (H3G34) DHGs. II. To correlate argininosuccinate synthase 1 (ASS1) and arginase tumor expression and Cerebral spinal fluid (CSF)/systemic arginine levels with survival.

III. To correlate levels of cell free DNA and other liquid biomarkers in the context of imaging response criteria and clinical outcome.

IV. To assess the microbiome in the context of imaging response criteria and clinical outcome.

V. To describe the pharmacokinetics of ADI-PEG 20 in combination with radiotherapy and TMZ and in maintenance treatment in children, adolescent and young adults with HGG.

VI. To describe the pharmacodynamics of ADI-PEG 20 in combination with radiotherapy and TMZ and in maintenance treatment in children, adolescent and young adults with HGG.

VII. To assess immunogenicity of ADI-PEG 20 in combination with radiotherapy and TMZ and in maintenance treatment in children, adolescent and young adults with HGG.

VIII. To explore the use of serial single voxel magnetic resonance (MR) spectroscopy to evaluate on-target tumor metabolic changes with the use of ADI-PEG 20.

IX. To explore sex differences in arginine metabolism in participants with newly diagnosed high-grade glioma pre and post treatment with ADI-PEG 20.

X. To characterize immune micro-environment of tumor edge in comparison to tumor core. Inclusion of normal/reactive brain tissue will be used to compare baseline reactive transcriptional signature, including immune pathways activated in peritumoral regions of the brain.

OUTLINE: Participants will be enrolled into Phase 1 (dose escalation) where the pediatric RP2D of ADI-PEG 20 in combination with radiotherapy and daily TMZ (DLT period 1) as well as ADI-PEG 20 with TMZ during maintenance (DLT period 2) will be determined through a rolling-6 design and then followed by a planned Phase 2. Participants in Phase 2 will further be analyzed by cohort based on confirmed diagnosis of the following expressed biomarkers:

Cohort 1: Participants with newly diagnosed histone wild type (WT) HGG. (N=25).

Cohort 2: Participants with newly diagnosed H3K27 altered diffuse midline gliomas (DMG). (N=30).

Cohort 3: Participants with newly diagnosed H3G34 mutant diffuse hemispheric gliomas (DHG). (N=18).

Participants can receive treatment up to 104 weeks. After completing the 30-day toxicity evaluation period, participants will enter follow-up and additional follow-up data will be documented under the Pediatric Neuro-oncology Consortium (PNOC) COMP protocol. Participants will be followed under the PNOC COMP protocol until death or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically and molecularly confirmed newly diagnosed World Health Organization (WHO) grade 3 or 4 glioma.

   1. Phase 1: any newly diagnosed HGG (including DMG of any location and primary spinal cord tumors).
   2. Phase 2:

      * Cohort 1: Newly diagnosed non-pontine, non-spinal cord HGG histone-wildtype.
      * Cohort 2: Newly diagnosed non-pontine, non-spinal cord H3K27 altered diffuse midline glioma (DMG).
      * Cohort 3: Newly diagnosed non-pontine, non-spinal cord H3G34 mutant diffuse hemispheric glioma (DHG).
2. Prior surgery: must have undergone maximal safe resection. For patients with DMG of the pons, biopsy is sufficient.
3. Prior Therapy: Participants must NOT have received ANY prior therapy (except surgery) before enrollment on study.
4. Tumor Tissue Requirement: Participants must have sufficient tumor tissue (5-10 unstained formalin-fixed paraffin-embedded (FFPE) slides or a tumor block) for study enrollment.
5. Age:

   Phase 1:

   o 3 to <18 years of age.

   Phase 2:
   * Cohort 1: 3 to 25 years of age.
   * Cohorts 2 & 3: 3 to 39 years of age.
6. Performance Score: Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants <=16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. Corticosteroids: Participants who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
8. Organ Function Requirements:

   1. Peripheral absolute neutrophil count (ANC) >= 1000/mm^3.
   2. Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
   3. Creatinine Clearance (CrCl) or estimated glomerular filtration rate (eGFR) with cutoff value of ≥ 60 mL/min for renal function in participants with age ≥ 18 years. For participants < 18 years old, estimate eGFR using the Schwartz equation. eGFR (mL/min/1.73 m^2) = (k × Height (cm)) / Serum Creatinine (mg/dL).
   4. Total bilirubin <= 1.5 x upper limit of normal (ULN) for age; in presence of Gilbert's syndrome, total bilirubin < 3 x ULN or direct bilirubin < 1.5 x ULN.
   5. alanine aminotransferase (ALT) <= 3 x ULN.
   6. aspartate aminotransferase (AST) <= 3 x ULN.
   7. Participants with seizure disorder may be enrolled if well controlled. Participants on non-enzyme inducing anticonvulsants may be excluded pending interaction(s) with study drug.
9. The effects of ADI-PEG 20 have been shown to be associated with embryofetal toxicity in rodents. For this reason and because chemotherapy used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. A legal parent/guardian or participant must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.
11. Participants must enroll on PNOC COMP if PNOC COMP is open to accrual at the enrolling institution.

Exclusion Criteria:

1. Participants who have received any systemic therapy or RT, including any investigational agents.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ADI-PEG 20 such as pegylated compounds.
3. Phase 2 cohorts: tumors with epicenter in pons or spinal cord
4. Participants with metastatic or leptomeningeal disease. Multi-focal disease should be discussed with the study chairs,
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection that would interfere with the study.
6. Women of childbearing potential must not be pregnant or breast-feeding.
7. Human immunodeficiency virus (HIV)-positive participants will be ineligible if HIV therapy regimen has not been stable for at least 4 weeks or there is intent to change the regimen within 8 weeks following enrollment, or if they are severely immunocompromised.
8. Corrected QT Interval (QTc) cutoff >480 ms.

Important note: The eligibility criteria listed above are interpreted literally and cannot be waived.

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2032-06-30 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Treatment-emergent Adverse Events (TrAE) (Phase 1) | Up to 104 weeks
  Proportion of participants in Phase 1 with treatment-emergent adverse events as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) will be reported.
Progression-Free Survival (PFS) for HGG histone-WT (Phase 2, Cohort 1) | Up to 12 months
  PFS for participants in Phase 2, Cohort 1 is defined as the median number of days participants remained progression free at 12 months. Participants without a documented tumor progression or death will be censored on the date of their last evaluable tumor assessment. Participants without a documented tumor progression or death before initiation of another anti-tumor therapy will be censored on the date of their last evaluable tumor assessment prior to or on the date of the new anti-tumor therapy. PFS estimates will be obtained from the Kaplan-Meier curve. An appropriate variance term that accounts for censoring Greenwood's formula) will be used to construct the 95% confidence intervals.
Progression-Free Survival (PFS) for H3K27 altered diffuse midline glioma (DMG) (Phase 2, Cohort 2) | Up to 12 months
  PFS for participants in Phase 2, Cohort 2 is defined as the median number of days participants remained progression free at 12 months. Participants without a documented tumor progression or death will be censored on the date of their last evaluable tumor assessment. Participants without a documented tumor progression or death before initiation of another anti-tumor therapy will be censored on the date of their last evaluable tumor assessment prior to or on the date of the new anti-tumor therapy. PFS estimates will be obtained from the Kaplan-Meier curve. An appropriate variance term that accounts for censoring Greenwood's formula) will be used to construct the 95% confidence intervals.
Progression-Free Survival (PFS) for H3G34 mutant diffuse hemispheric glioma (DHG) (Phase 2, Cohort 3) | Up to 10 months
  PFS for participants in Phase 2, Cohort 3 is defined as the median number of days participants remained progression free at 10 months. Participants without a documented tumor progression or death will be censored on the date of their last evaluable tumor assessment. Participants without a documented tumor progression or death before initiation of another anti-tumor therapy will be censored on the date of their last evaluable tumor assessment prior to or on the date of the new anti-tumor therapy. PFS estimates will be obtained from the Kaplan-Meier curve. An appropriate variance term that accounts for censoring Greenwood's formula) will be used to construct the 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco; Tom Davidson, MD, Study Chair — Children's Hospital Los Angeles
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be shared with study collaborators during the course of the study.